CLINICAL TRIAL: NCT04111419
Title: Intensive Management of Blood Pressure and Cholesterol in Elderly Chinese With Hypertension and Atrial Fibrillation (IMPRESSION)
Brief Title: Intensive Management of Blood Pressure and Cholesterol in Elderly Chinese With Hypertension and Atrial Fibrillation
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPRESSION
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation; Hypertension
Keywords: intensive management; blood pressure; blood cholesterol
MeSH Terms: conditions — Atrial Fibrillation; Hypertension | interventions — Amlodipine; Atorvastatin; allisartan isoproxil

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly divided into four groups, taking amlodipine/atorvastatin (5/10mg tablet) once a day or amlodipine/atorvastatin (5/20mg tablet) once a day or amlodipine/atorvastatin (5/10mg tablet)+allisartan (240mg/tablet) once a day or amlodipine/atorvastatin (5/20mg tablet)+allisartan (240mg/tablet) once a day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intensive blood pressure and cholesterol control (Experimental)
  Interventions: Drug: Amlodipine/Atorvastatin 5 Mg-20 Mg ORAL TABLET; Drug: Allisartan Isoproxil
- Intensive blood pressure and routine cholesterol control (Active Comparator)
  Interventions: Drug: Amlodipine/Atorvastatin 5 Mg-10 Mg ORAL TABLET; Drug: Allisartan Isoproxil
- Routine blood pressure and intensive cholesterol control (Active Comparator)
  Interventions: Drug: Amlodipine/Atorvastatin 5 Mg-20 Mg ORAL TABLET
- Routine blood pressure and cholesterol control (Active Comparator)
  Interventions: Drug: Amlodipine/Atorvastatin 5 Mg-10 Mg ORAL TABLET

INTERVENTIONS:
Drug: Amlodipine/Atorvastatin 5 Mg-20 Mg ORAL TABLET — amlodipine/atorvastatin (5/20mg tablet) once a day
  Arms: Intensive blood pressure and cholesterol control; Routine blood pressure and intensive cholesterol control
Drug: Amlodipine/Atorvastatin 5 Mg-10 Mg ORAL TABLET — amlodipine/atorvastatin (5/10mg tablet) once a day
  Arms: Intensive blood pressure and routine cholesterol control; Routine blood pressure and cholesterol control
Drug: Allisartan Isoproxil — allisartan (240mg/tablet) once a day
  Arms: Intensive blood pressure and cholesterol control; Intensive blood pressure and routine cholesterol control

SUMMARY:
1. Study name: Intensive management of blood pressure and cholesterol in elderly Chinese with hypertension and atrial fibrillation (IMPRESSION)
2. Medicine: amlodipine/atorvastatin (5/10mg tablet); amlodipine/atorvastatin (5/20mg tablet); allisartan (240mg/tablet).
3. Rationale: controlling blood pressure and cholesterol are both effective means to reduce cardiovascular risks, however, it is still unknown whether high cardiovascular risk patients with atrial fibrillation would benefit from intensive management of blood pressure and cholesterol.
4. Objective: To evaluate the efficacy and safety of intensive management of blood pressure and cholesterol.
5. Study design: This study is a multi-center, randomized and controlled clinical trial with four equally sized treatment groups: amlodipine/atorvastatin (5/10mg tablet); amlodipine/atorvastatin (5/20mg tablet); amlodipine/atorvastatin (5/10mg tablet)+allisartan (240mg/tablet); amlodipine/atorvastatin (5/20mg tablet)+allisartan (240mg/tablet).
6. Study population: Men and Women aged over 65 years (n=1200) meeting the inclusion/exclusion criteria.
7. Randomization and treatment: After stratification by centers, eligible patients will be randomly divided into four groups, taking amlodipine/atorvastatin (5/10mg tablet) once a day or amlodipine/atorvastatin (5/20mg tablet) once a day or amlodipine/atorvastatin (5/10mg tablet)+allisartan (240mg/tablet) once a day or amlodipine/atorvastatin (5/20mg tablet)+allisartan (240mg/tablet) once a day.
8. Follow up: 3 years.
9. Sample size: a total of 1200 patients should be enrolled in the combination.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in September 2019, recruitment will start. Patients enrollment will be performed between November 2019 to November 2020. All patients should be followed up before December 2023.

DETAILED DESCRIPTION:
1. Study name: Intensive management of blood pressure and cholesterol in elderly Chinese with hypertension and atrial fibrillation (IMPRESSION)
2. Medicine: amlodipine/atorvastatin (5/10mg tablet); amlodipine/atorvastatin (5/20mg tablet); allisartan (240mg/tablet).
3. Rationale: controlling blood pressure and cholesterol are both effective means to reduce cardiovascular risks, however, it is still unknown whether high cardiovascular risk patients with atrial fibrillation would benefit from intensive management of blood pressure and cholesterol.
4. Objective: To evaluate the efficacy and safety of intensive management of blood pressure and cholesterol, especially in hypertensive patients with atrial fibrillation.
5. Study design: This study is a multi-center, randomized and controlled clinical trial with four equally sized treatment groups: amlodipine/atorvastatin (5/10mg tablet); amlodipine/atorvastatin (5/20mg tablet); amlodipine/atorvastatin (5/10mg tablet)+allisartan (240mg/tablet); amlodipine/atorvastatin (5/20mg tablet)+allisartan (240mg/tablet).
6. Study population: Men or women aged over 65 years (n=1200) will be screened for atrial fibrillation. Atrial fibrillation patients who never took antihypertensive drugs or stop antihypertensive drugs for more than 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg or who is on monotherapy for at least 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg will be recruited. Before randomization, two visits should be performed and 6 clinic blood pressures should be recorded. The average of the 6 clinic blood pressures should be 140-179 mmHg in systolic and/or 90-109 mmHg in diastolic. Regardless of whether the office blood pressure meets the enrollment conditions, a one-week home blood pressure measurement should be performed before randomization. Patient should sign the written consent form before screening and be able to go to the clinic by him/herself. Exclusion criteria included: suspected or confirmed secondary hypertension; history of coronary heart disease, myocardial infarction, heart failure, stroke or dementia; taking other drugs that might affect blood pressure; liver dysfunction, serum creatinine ≥1.5 mg/dL (133 μmol/L), urine protein positive; serum potassium >5.0 mmol/L or <3.5 mmol/L; uncontrolled diabetes (HbA1c >8%); BMI ≥35kg/m²; elderly care patients; or patients who are participating in other clinical trials.
7. Randomization and treatment: After stratification by centers, eligible patients will be randomly divided into four groups, taking amlodipine (5 mg/tablet)+ once a day or amlodipine besylate tablets (5 mg/tablet) + hydrochlorothiazide tablets (25 mg/tablet) once a day.
8. Follow up: Sitting office blood pressures and electrocardiogram should measured by an OMRON device. Medical history should be recorded. Clinical examinations including home blood pressure, electrocardiogram, blood and urine routine tests and biochemical tests should be performed. Patients should be followed up every three months. Before the follow-up, patients should perform a one-week home blood pressure monitoring.
9. Sample size and statistical analysis: At least 300 eligible patients should be enrolled in each group, and a total of 1200 patients should be enrolled in total. Data will be analyzed by using the SAS software. ANOVA will be used to compare the parameters between groups and the difference between the four groups with the calculation of 95% confidence interval. In addition, a covariance analysis will also be used in the analysis of baseline parameters.
10. Timeline: After obtaining the approval of Ethics Committee of Ruijin Hospital in September 2019, recruitment will start. Patients enrollment will be performed between October 2019 to October 2020. All patients should be followed up before December 2023. Database construction and statistical analysis will be conducted at the same time, appropriate domestic and international conferences will be selected to publish the research results. The main results will be published in international professional medical journals.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

Men or women aged over 65 years. patients who never took antihypertensive drugs or stop antihypertensive drugs for more than 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg or who is on monotherapy for at least 2 weeks with systolic blood pressure of 140-179 mmHg and / or diastolic blood pressure of 90-109 mmHg.

Patient who sign the written consent and are able to go to the clinic by him/herself.

Exclusion Criteria:

suspected or confirmed secondary hypertension; taking two or more antihypertensive drugs; patients who never take antihypertensive drugs with a clinic blood pressure over 180/110 mmHg or treated patients with a clinic blood pressure over 160/100 mmHg or patients with a home blood pressure below 130/80 mmHg; history of coronary heart disease, myocardial infarction, heart failure, stroke or dementia; taking other drugs that might affect blood pressure; liver dysfunction, serum creatinine ≥1.5 mg/dL (133 μmol/L), urine protein positive; serum potassium >5.0 mmol/L or <3.5 mmol/L; uncontrolled diabetes (HbA1c >8%); BMI ≥35kg/m²; severe OSAS; patients who are participating in other clinical trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Combined cardiovascular end-point events | 3 years
  Fatal and non-fatal stroke, acute MI and cardiovascular death

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China